CLINICAL TRIAL: NCT02296489
Title: An Association Between Asthma Severity and Capnography Parameters
Status: Completed | Type: Observational
Sponsor: Oridion (Industry)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: D007773
Record Dates: First submitted 2014-11-04; First posted 2014-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
  Interventions: Device: Capnostream20p
- Asthma patients
  Interventions: Device: Capnostream20p

INTERVENTIONS:
Device: Capnostream20p — The device will be used to monitor respiratory co2 values during the methacholine challenge, a well known diagnostic procedure

SUMMARY:
Asthma is a common chronic disorder of the airways characterized by periods of reversible airflow obstruction known as asthma episodes or attacks. Asthma attacks are caused by chronically hyperactive (contraction of the muscles surrounding the airways) and inflamed airways, leading to airflow obstruction, and may be mild, moderate, or severe enough to become life-threatening events. Severity of asthma exacerbation is assessed through medical history and lung function measurements with Spirometer and requires full cooperation of the patient. Thus, in uncooperative populations or during emergency medical situations the spirometer cannot be used. As an alternative, capnography data has been proposed as an indicator of bronchospasm in asthma. Previous studies found correlations between the capnography parameters and methacholine challenge in asthma patients. However, the relationship between capnography parameters and severity of asthma or severity of asthma exacerbation have not been well characterized. The study hypothesis is that within the clinical population that is invited to do the methacholine challenge, a different waveform pattern in asthma patients will be detected and possibly a correlation between the severity of obstruction and pattern of waveform during the methacholine challenge. In this proposed feasibility observational study, sixty subjects, both men and women, who will be invited to participate in the methacholine challenge in the Institute of Pulmonary Medicine at Rabin Medical Center, will be recruited to the study. Respiratory information will be recorded using the CapnostreamTM20p while the subjects will wear the non-invasive Smart CapnoLine® Plus sampling line. Additionally, FeNO will be measured using a DENOX 88 device during the methacholine challenge.

ELIGIBILITY:
Inclusion Criteria:

1. The subject was invited to participate in methacholine challenge for the purposes of clinical assessment, with no relation to this study
2. Age 18-70
3. Ability to sign informed consent form

Exclusion Criteria:

1. Cannot or not willing to have capnography measurement during the entire methacholine challenge
2. Has or had in the past chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty subjects, both men and women, who will be invited to participate in the methacholine challenge in the Institute of Pulmonary Medicine at Rabin Medical Center, regardless to the study, will be recruitment to the study.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measuring the change in expired CO2 over time in asthma patients during the methacholine challenge. | 1 year

SECONDARY OUTCOMES:
Finding a correlation between the change in expired CO2 and the severity of asthma as reflected by PC20. | 1 year
Finding a correlation between the change in expired CO2 and the severity of asthma as reflected by the frequency of symptoms according the Asthma Severity Tool (AST). | 1 year
Finding correlations between changes in capnography parameters and the severity of asthma as reflected by preliminary FEV1, forced vital capacity (FVC), FEV1/FVC, and peak expiratory flow rate. | 1 year
Finding a correlation between change in expired CO2 and fraction of exhaled nitric oxide (FeNO). | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Institute Rabin Medical center, Beilinson Hospital, Petah Tikva, Israel